CLINICAL TRIAL: NCT03295825
Title: Prospective Multi-centre Clinical Study to Assess the Clinical Validity of the Heparin Binding Protein Assay to Indicate the Presence and Outcome of Sepsis in Patients With Suspected Infection Following Emergency Department Admission
Brief Title: Heparin Binding Protein in Early Sepsis Diagnosis
Acronym: PROMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROMPT
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Sepsis; Infection
Keywords: Heparin binding protein; Mortality
MeSH Terms: conditions — Sepsis; Infections | interventions — Environmental Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biomarker (Other): Blood sampling
  Interventions: Diagnostic Test: Biomarker

INTERVENTIONS:
Diagnostic Test: Biomarker — Measument of heparin-binding protein in the serum of patients
  Other Names: Heparin Binding Protein

SUMMARY:
The primary objective of this study is to use heparin-binding protein (HBP) concentration to indicate the presence, or outcome, of sepsis over 72 hours after ED admission. The secondary objectives of this study are to separately evaluate the performance of HBP to predict outcome in patients with suspected infection over 12-24 hours after ED admission.

DETAILED DESCRIPTION:
The purpose of this prospective, non-interventional, multi-centre clinical study is to assess the clinical validity of the Heparin Binding Protein (HBP) assay for indicating the presence, or outcome, of severe sepsis (including septic shock), over 72 hours, in patients with suspected infection following emergency department admission.

Sepsis is an increasingly common cause of morbidity and mortality, with approximately 150,000 people in Europe and 215,000 people in the US dying of severe sepsis each year. Deaths attributable to sepsis continue to rise due to an increase in incidence of the disease, which can be attributed to numerous factors including the aging population, the increased number of immuno-compromised patients, the increased use of invasive surgery and the increased incidence of microbial resistance.

The sepsis syndrome was first described in the 1992 publication by Bone et al detailing the conclusions of the ACCP/SCCM Consensus Conference held in 1991, which first introduced the Systemic Inflammatory Response Syndrome (SIRS) classification system. Systemic Inflammatory Response Syndrome (SIRS) is considered to be present when patients have 2 or more of the following clinical findings:

* body temperature, >38ºC or <36ºC
* heart rate, >90 beats per minute
* respiratory rate of >20 breaths per minute or a PaCO2 of <32mm Hg
* white cell count of >12,000 cells per µL or <4,000 per µL, or >10% immature (band) forms According to the suggested definitions, sepsis is defined as SIRS plus confirmed infection, severe sepsis is defined as sepsis associated with organ dysfunction, hypoperfusion, or hypotension and septic shock is defined as sepsis-induced hypotension, persisting despite adequate fluid resuscitation.

Diagnosis of sepsis traditionally relies on identification of the above symptoms, as well as culturing techniques to confirm and identify the infection. This method of diagnosis is, however, far from ideal as it has been demonstrated that SIRS criteria are poorly predictive of subsequent events in the sepsis cascade and that approximately one half of severe sepsis cases are culture negative. In addition, the assay time for culture-based diagnosis is 24 to 48 hours, where it has been shown that diagnosis of severe sepsis and septic shock as early as possible is important, as each hour of delay in effective antimicrobial administration is associated with an average decrease in survival of 7.6%. Although the majority of severe sepsis patients receive treatment in an intensive care unit (ICU), it is estimated that up to two thirds of those patients initially present to the emergency department (ED), and that approximately 20% of patients with confirmed infection who present to the ED with uncomplicated sepsis progress to severe sepsis or septic shock within 72 hours.

This high incidence of early progression to severe sepsis and septic shock among patients presenting to the ED highlights the time-sensitive nature of diagnosis, especially in patients who initially do not appear critically ill. Therefore early intervention to prevent subsequent or worsening clinical deterioration is key to the successful treatment of patients. However, two major impediments to the effectiveness of sepsis treatment strategies are a failure to recognise the early stages of the disease and underestimation of its severity, as it is difficult to determine which of the patients with signs of infection on initial evaluation have, or will develop, more serious illness. Several outcome prediction models, including Acute Physiology and Chronic Health Evaluation (APACHE) IV, the Simplified Acute Physiology Score (SAPS) III, the Logistic Organ Dysfunction Score (LODS), and the Mortality Probability Model (MPM) III have therefore been developed for use in clinical practice. Moreover patients admitted in the ED with at least two of three clinical signs (hypotension, tachypnea, altered mental status) are highly possible to suffer from sepsis. These three clinical signs are the qSOFA score. Data from the Hellenic Sepsis Study Group put into question if the qSOFA score can predict sepsis in the ED with sensitivity that exceeds 65% (15, 16). There is, therefore, still an unmet need for a diagnostic tool that can identify those patients at risk of developing more severe disease, and although a number of laboratory measures or novel sepsis biomarkers have been proposed for clinical use, there is currently no single accepted biomarker or combination of biomarkers for use in patients with suspected sepsis.

The recent publication by Linder et al(17) has shown that measurement of heparin binding protein (HBP), also known as azurocidin or CAP37, in febrile patients presenting to the ED shows a close correlation between increased plasma HBP levels and the development of severe sepsis with hypotension or shock. In this prospective study of 233 febrile adult patients with suspected infection, 26 were diagnosed with severe sepsis with septic shock, 44 with severe sepsis without septic shock, 100 with sepsis, 43 with infection without SIRS and 20 with SIRS without infection. Using a cut-off of 15ng/mL, HBP showed a sensitivity in diagnosing severe sepsis (with or without septic shock) of 87.1%, a specificity of 95.1%, a positive predictive value (PPV) of 88.4% and a negative predictive value (NPV) of 94.5%, which exceeded those values obtained for the other tested markers. Receiver-operating characteristic (ROC) curves also demonstrated that HBP was the best predictor of severe sepsis, with an area under the curve (AUC) value of 0.95. It is therefore hypothesised that HBP may be used for the early identification of patients at risk of developing severe sepsis and septic shock. In addition, it was observed that 20 of the patients with severe sepsis were monitored with serial plasma sample collection during the course of the disease, and that the 18 of these patients who survived had HBP levels that decreased rapidly when the clinical signs improved and the blood pressures were normalised. It is therefore further hypothesised that a decrease in HBP levels may be used to predict survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Male or female
* Written informed consent
* Suspected infection
* Presence of at least ONE of the following:

Temperature > 38°C Temperature < 36°C Heart rate > 90 bpm Respiratory rate > 20/min Self reported fever/chills

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
ΗΒΡ for sepsis diagnosis | 72 hours
  Sensitivity of ΗΒΡ for sepsis diagnosis. Every value over 90% is considered satisfactory.

SECONDARY OUTCOMES:
Diagnostic performance of HBP for sepsis | 72 hours
  Specificity, positive predictive value and negative predictive value of HBP to diagnose sepsis
Diagnostic performance of HBP for septic shock | 72 hours
  Specificity, positive predictive value and negative predictive value of HBP to diagnose septic shock
Diagnostic performance of HBP for early death | 72 hours
  Sensitivity, specificity, positive predictive value and negative predictive value of HBP to predict unfavorable outcome
Diagnostic performance of HBP for death | 28 days
  Sensitivity, specificity, positive predictive value and negative predictive value of HBP to predict unfavorable outcome

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Giamarellos-Bourboulis, MD, PhD, Study Chair — National and Kapodistrian University of Athens
Locations (6):
- Greece (6):
  - Nafplion General Hospital, Nafplion, Argos
  - 4th Department of Internal Medicine, ATTIKON University Hospital, Athens, Attica
  - Department of Internal Medicine, Chalkida General Hospital, Chalcis
  - Department of Internal Medicine, Siros General Hospital, Ermoupoli
  - Department of Internal Medicine, Sparti General Hospital, Sparti
  - 2nd Department of Surgery, G.Gennimatas Thessaloniki General Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linder A, Christensson B, Herwald H, Bjorck L, Akesson P. Heparin-binding protein: an early marker of circulatory failure in sepsis. Clin Infect Dis. 2009 Oct 1;49(7):1044-50. doi: 10.1086/605563. PMID 19725785
- [Derived] Safarika A, Wacker JW, Katsaros K, Solomonidi N, Giannikopoulos G, Kotsaki A, Koutelidakis IM, Coyle SM, Cheng HK, Liesenfeld O, Sweeney TE, Giamarellos-Bourboulis EJ. A 29-mRNA host response test from blood accurately distinguishes bacterial and viral infections among emergency department patients. Intensive Care Med Exp. 2021 Jun 18;9(1):31. doi: 10.1186/s40635-021-00394-8. PMID 34142256